CLINICAL TRIAL: NCT05194878
Title: Phase III Study of Neoadjuvant FOLFOXIRI Chemotherapy Versus Immediate Surgery for High-risk Resectable Stage II and III Colon Cancers
Brief Title: Neoadjuvant FOLFOXIRI Versus Immediate Surgery for Stage II and III Colon Cancers
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Pei-Rong Ding, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-FXY-244
Record Dates: First submitted 2021-12-21; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Colon Cancer Stage II; Colon Cancer Stage III
Keywords: neoadjuvent chemotherapy; FOLFOXIRI; colon caner
MeSH Terms: conditions — Colonic Neoplasms | interventions — Colectomy; Chemotherapy, Adjuvant; Folfox protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant chemotherapy (Experimental): 12 weeks of FOLFOXIRI neuoadjuvantly followed by surgery and adjuvant chemotherapy
  Interventions: Drug: neoadjuvant chemotherapyI; Procedure: Colectomy
- Postoperative chemotherapy (Active Comparator): surgery followed by 24 weeks of FOLFOX or CapeOX or Cape
  Interventions: Procedure: Colectomy; Drug: adjuvant chemotherapy

INTERVENTIONS:
Drug: neoadjuvant chemotherapyI — mFOLFOXIRI (IV oxaliplatin given over 120 min at a dose of 85 mg/m2 on day 1 followed by IV leucovorin 400 mg/m2 over 2h, IV Irinotecan 150 mg/m2 and IV infusional 5-Fluorouracil 2400 mg/m2 over 48h every 14 days) for 6 cycles followed by colectomy (3 to 6 weeks after) . If PD was observed after 3 cycles, direct colectomy was performed.
  Other Names: mFOLFOXIR
  Arms: Neoadjuvant chemotherapy
Procedure: Colectomy — Radical colectomy
Drug: adjuvant chemotherapy — mFOLFOX6 (IV oxaliplatin given over 120 min at a dose of 85 mg/m2 on day 1 followed by IV leucovorin 400 mg/m2 over 2h, IV bolus 5-Fluorouracil 400 mg/m2 and IV infusional 5-Fluorouracil 2400 mg/m2 over 46h every 14 days) . CAPOX (IV oxaliplatin given over 120 min at a dose of 130 mg/m2 on day 1, oral capecitabine 1000 mg/m2 twice daily on days 1 through 14 every 21 days) . Oral capecitabine 1000 mg/m2 twice daily on days 1 through 14 every 21 days. The plan and cycles are determined according to the surgical pathology and physical conditions.
  Other Names: FOLFOX/CapeOX/Cape
  Arms: Postoperative chemotherapy

SUMMARY:
BACKGROUND:

In patients with high risk stage II and stage III colon cancer (CC), curative surgery followed by adjuvant chemotherapy with FOLFOX or CAPOX regimens has become a standard treatment. However, 20 to 30 % of these patients will develop distant metastasis, which ultimately result in death. Perioperative chemotherapy is a promising strategy with potential benefits that could be more effective at eradicating micrometastases. Moreover, shrinking tumor before surgery not only facilitate removal of all the tumor by the surgeon but also reduce tumor cell spreading during the procedure. With recent advances in radiology, preoperative computed tomography allows a good prediction of tumor stage (wall penetration and nodal involvement) prior to surgery. The investigators conducted the present randomized study to explore whether perioperative chemotherapy with FOLFOXIRI regimen compared with postoperative chemotherapy could improve disease-free survival in patients with radiologically staged, High-risk, but resectable Stage II or III colon cancer.

OBJECTIVE:

The primary objective of this study is to evaluate the efficacy of perioperative chemotherapy with FOLFOXIRI regimen compared to postoperative chemotherapy in patients with High-risk Resectable Stage II and III colon cancer. Secondary objectives are efficacy in terms of R0 resection rate, overall survival (OS), relapse-free survival (RFS), down-staging of primary tumors, and tolerability of perioperative therapy and postoperative complications.

DETAILED DESCRIPTION:
This trial is a a two-arm, multicenter, open labelled, prospective, randomized phase III studies. Eligible patients with High-risk Resectable Stage II and III (T4 or T3 with extramural depth≧5 mm) colon cancer patients will be randomly assigned, in a 2:1 ratio, to receive either perioperative or postoperative chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma or high grade dysplasia on histology plus unequivocal radiological evidence of invasive cancer of the colon(≥ 12 cm from the anal verge).
* pMMR in immunohistochemical detection or MSI-H in MSI test.
* Determined preoperatively by either spiral or multidetector CT: high risk T3 (tumor disruption of muscle wall and extension into pericolic fat with more than 5 mm protrusion into adjacent mesenteric fat) or T4 (tumor penetrates to the surface of the visceral peritoneum or directly invades or is adherent to adjacent organs or structures).
* Patients presenting with acute colonic obstruction may enter the trial only after obstruction is relieved by a successful defunctioning stoma, and when recovered to a fitness level consistent with the other eligibility criteria
* Adequate full blood count: WBC >3.0 x109/l; Plts >100 x109/l. Anaemia (Hb < 10.0 g/dl) is not an exclusion, but should be corrected by transfusion prior to surgery and chemotherapy. If Hb remains low despite transfusions, surgery and chemotherapy can be given at the decision of the surgical and oncology teams.
* Adequate renal biochemistry: serum creatinine was less than 1.5 times the normal value.
* Adequate hepatobiliary function: serum total bilirubin and ALT were less than 1.5 times the normal value.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* Any patient for whom radiotherapy is advised by the MDT
* Strong evidence of distant metastases or peritoneal nodules (M1)
* dMMR in immunohistochemical detection or MSI-L/MS-S in MSI test.
* Peritonitis (secondary to perforated tumour)
* Colonic obstruction that has not been defunctioned
* Serious medical comorbidity, eg uncontrolled inflammatory bowel disease, uncontrolled angina or recent (<6 months) MI
* Another serious medical condition judged to compromise ability to tolerate neoadjuvant therapy and/or surgery
* Any other malignant disease within the preceding 5 years with the exception of non-melanomatous skin cancer, carcinoma in situ and early stage disease with a recurrence risk <5%

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 2 years
  Defined as the time from randomization to relapse or death, whichever occurred first

SECONDARY OUTCOMES:
Overall survival | 5 years
  Defined as the time from randomization to death from any cause
Down-staging of primary tumors | 1 year
  Down-staging of the resected tumour as measured by histopathological tumour diameter and stage according to the TNM staging system of AJCC (7th version)
Chemotherapy toxicity | through chemotherapy administration, up to 6 months
  The grade of toxicity will be assessed using the NCI common toxicity criteria, version 4.0
R0 resection rate | after surgery completed, up to 1 month
  Quality of resection specimen
Surgical morbidity | 30 days post surgery
  Complication after surgery
CT staging | from randomization to surgery completed, up to 6 months
  the accuracy of CT staging
CT assessment of response to neoadjuvant treatment | up to 6 months
  CT evaluation of the thickness of tumor walls or tumor diameter or tumor length. Efficacy evaluation will be assessed using the RECIST criteria, version 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- 651 Dongfeng Road East, Guangzhou, Guangdong, China